CLINICAL TRIAL: NCT00865501
Title: Importance of Aldosterone in the Pathogenesis of Hypertensive Heart Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFO-TP5-I
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Primary Hypertension
Keywords: primary hypertension; aldosterone; left ventricular hypertrophy
MeSH Terms: conditions — Essential Hypertension; Hypertrophy, Left Ventricular | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): spironolactone
  Interventions: Drug: spironolactone
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: spironolactone — 25mg per oral once daily
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The Renin-Angiotensin-Aldosterone-system is important in the development of cardiovascular organ damage caused by arterial hypertension. This study aims at evaluating the importance of aldosterone with regard to hypertension induced damage to the heart. In order to do this the investigators will perform a comparative cross-sectional study in hypertensives and normotensives. In addition as interventional part the hypertensives will be treated with a mineralocorticoid-receptor blocker (spironolactone).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis hypertension (BP higher than 139/89)

Exclusion Criteria:

* Antihypertensive pretreatment
* Contraindications against spironolactone
* Being unable to understand or comply with study procedures

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
left ventricular mass | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, FACP, Principal Investigator — Universität Erlangen-Nurnberg
Locations (1):
- University Erlangen-Nürnberg, Nephrology and Hypertension, Erlangen, Germany